CLINICAL TRIAL: NCT04911192
Title: Catheter-Directed Pulmonary Re Perfusion in Treatment of Intermediate and High Risk Pulmonary Embolism Patients and Its Impact on Pulmonary Artery Pressure
Brief Title: Catheter-Directed Pulmonary Reperfusion in Treatment of Pulmonary Embolism Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliaa Salama Ahmed Omar, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR in PE
Record Dates: First submitted 2021-05-25; First posted 2021-06-02 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- systemic thrombolysis group (No Intervention): patients without any contraindications for systemic fibrinolytic therapy will be treated with traditional systemic thrombolysis (intravenous administration of streptokinase).
- mechanical fragmentation group (Active Comparator): patients will be treated with catheter-directed mechanical fragmentation under fluoroscopy guidance. This group will include patients with absolute contraindication for fibrinolytic therapy.
  Interventions: Procedure: mechanical fragmentation
- In Situ thrombolysis group (Active Comparator): patients will be treated with bed side administration of low dose of local thrombolytic therapy (In Situ) via a trans-Jugular Swan-Ganz pulmonary artery catheter. with guidance of the pressure waveforms obtained from SGC(Swan-Ganz pulmonary artery catheter) and echocardiography guidance for ideal Catheter placement. This group will include the patients with relative contraindications for systemic thrombolysis, contraindications for contrasted administration (patients with renal impairment) and also patients with contraindications for radiation exposure (pregnant women).
  Interventions: Procedure: In Situ thrombolysis

INTERVENTIONS:
Procedure: mechanical fragmentation — patients who will be treated with catheter-directed mechanical fragmentation under fluoroscopy guidance. This group will include patients with absolute contraindication for fibrinolytic therapy
  Arms: mechanical fragmentation group
Procedure: In Situ thrombolysis — Group (C) will include the patients who will be treated with bed side administration of low dose of local thrombolytic therapy (In Situ) via a trans-Jugular Swan-Ganz pulmonary artery catheter. with guidance of the pressure waveforms obtained from SGC (Swan-Ganz catheter) and echocardiography guidance for ideal Catheter placement. This group will include the patients with relative contraindications for systemic thrombolysis, contraindications for contrasted administration (patients with renal impairment) and also patients with contraindications for radiation exposure (pregnant women).
  Arms: In Situ thrombolysis group

SUMMARY:
* Primary objective: to evaluate the success and mortality rates of catheter-directed reperfusion therapy in comparison to traditional use of systemic intravenous fibrinolytic therapy, will focus at safety of such management measured by in-hospital mortality and prevalence of severe adverse events.
* Secondary objective: to assess the feasibility of catheter-directed reperfusion in management of intermediate and high risk pulmonary embolism in Assiut University hospital and its reflection on pulmonary artery pressure

DETAILED DESCRIPTION:
Venous thromboembolic disease represents one of the most important causes of cardiovascular death in the world. Symptomatic pulmonary embolism (PE) occurs in about 500,000 patients annually, with an estimated mortality as high as 30% in high-risk patients .

High-risk pulmonary embolism clinically manifests with hemodynamic instability and systemic hypotension (systolic blood pressure < 90 mm Hg, pressure drop of more than 40 mm Hg or requiring administration of inotropic agents. In this form of PE (pulmonary embolism) imaging studies usually reveal a "saddle embolus" at the bifurcation of the pulmonary trunk, embolism of the main pulmonary artery, or embolic occlusion of at least two lobar arteries.

Mortality in high-risk pulmonary embolism is at the level of 60%, and in 66% of these patients fatal outcomes take place during the first hours from the onset of clinical symptoms. The remaining patients with severe pulmonary embolism , those with intermediate risk of mortality, do not reveal hypotension, but present with clinical symptoms comprising dyspnea and/or tachycardia. Estimated 30-day mortality in patients with intermediate risk PE (pulmonary embolism) is at the level of 15-20%, and these patients are at a risk of developing pulmonary hypertension and right ventricle heart failure. Given the fact that 40% of patients with class 4 or 5 of the Pulmonary Embolism Severity Index present with contraindications for systemic fibrinolytic therapy, Catheter-directed reperfusion therapy seems to be a promising alternative treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Both gender males and females.
* Patients with angiographically confirmed acute high risk pulmonary embolism with shock index >1.
* pulmonary arterial occlusion with >50% involvement of the central (main and/or lobar) pulmonary, and dysfunction of the right ventricle and elevated troponin.
* patients with high risk pulmonary embolism who remain unstable after receiving fibrinolysis
* patients with high risk PE pulmonary embolism who cannot receive fibrinolysis
* patients with intermediate high risk PE pulmonary embolism with adverse prognosis (new hemodynamic instability, worsening respiratory failure, severe RV (right ventricle) dysfunction, or major myocardial necrosis)

Exclusion Criteria:

* patients with echocardiographically confirmed right sided thrombi.
* patients with low-risk PE pulmonary embolism or submassive acute PE pulmonary embolism with minor RV (right ventricle) dysfunction, minor myocardial necrosis, and no clinical worsening
* Anaphylactic reaction to contrast media.
* Acute renal failure or severe chronic non-dialysis dependent kidney disease.
* Uncooperative patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of mortality (mortality rate) | 30-day
  number of deaths from total number of patients in each arm
Rate of complications | 7 days
  as major and minor bleedings
Rate of Success | 2 weeks
  number of cases with clinical success which defined as stabilization of hemodynamic parameters, resolution of hypoxia, survival from PE(pulmonary embolism) and restoring of right ventricular function (improvement of ghit ventricle and pulmonary artery pressure and decrease troponin level)

SECONDARY OUTCOMES:
Percent of Changes in mean blood pressure | Baseline (measured at first admission) and compared with measurements the following second, eighth, and 24th hours of the intervention.
  the percent of change in mean arterial blood pressure
Mean pulmonary artery pressure | Baseline (at addmission) and 24 hours after catheter-directed intervention
  Mean pulmonary artery pressure will be estimated by transthoracic echocardiography
Duration of ICU(intensive care unit) stay | "through study completion, an average of 1 year".
  the duration of ICU (intensive care unit) stay by days
Duration of hospital stay | "through study completion, an average of 1 year".
  the duration of hospital stay by days

CONTACTS AND LOCATIONS:
Overall Officials: mohamed M abd el hadi, prof, Principal Investigator — professor of chest diseases and tuberculosis; Ayman k hassan, lecturer, Study Director — Assiut University; olfat M El shinnawy, prof, Study Chair — Assiut University; Aliaa S Ahmed, MD, Principal Investigator — Assiut University

REFERENCES:
- [Background] Cohen AT, Agnelli G, Anderson FA, Arcelus JI, Bergqvist D, Brecht JG, Greer IA, Heit JA, Hutchinson JL, Kakkar AK, Mottier D, Oger E, Samama MM, Spannagl M; VTE Impact Assessment Group in Europe (VITAE). Venous thromboembolism (VTE) in Europe. The number of VTE events and associated morbidity and mortality. Thromb Haemost. 2007 Oct;98(4):756-64. doi: 10.1160/TH07-03-0212. PMID 17938798
- [Background] Goldhaber SZ, Visani L, De Rosa M. Acute pulmonary embolism: clinical outcomes in the International Cooperative Pulmonary Embolism Registry (ICOPER). Lancet. 1999 Apr 24;353(9162):1386-9. doi: 10.1016/s0140-6736(98)07534-5. PMID 10227218
- [Background] Nassiri N, Jain A, McPhee D, Mina B, Rosen RJ, Giangola G, Carroccio A, Green RM. Massive and submassive pulmonary embolism: experience with an algorithm for catheter-directed mechanical thrombectomy. Ann Vasc Surg. 2012 Jan;26(1):18-24. doi: 10.1016/j.avsg.2011.05.026. Epub 2011 Aug 31. PMID 21885244
- [Background] Anderson FA Jr, Zayaruzny M, Heit JA, Fidan D, Cohen AT. Estimated annual numbers of US acute-care hospital patients at risk for venous thromboembolism. Am J Hematol. 2007 Sep;82(9):777-82. doi: 10.1002/ajh.20983. PMID 17626254
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341